CLINICAL TRIAL: NCT02660671
Title: Behavioral Economic Approaches to Increase Colorectal Cancer Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 822504
Record Dates: First submitted 2016-01-19; First posted 2016-01-21 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Cancer of the Colon
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Usual care (Active Comparator): Email outreach
  Interventions: Behavioral: Email outreach
- Active choice (Experimental): Email outreach + active choice
  Interventions: Behavioral: Email outreach; Behavioral: Active choice
- Financial incentive + Active choice (Experimental): Email outreach + active choice + financial incentive
  Interventions: Behavioral: Email outreach; Behavioral: Active choice; Behavioral: Financial incentive

INTERVENTIONS:
Behavioral: Email outreach — Subjects will receive an email describing the importance of colorectal cancer screening and that s/he has been selected to participate in this VIP concierge service.
Behavioral: Active choice — S/he will receive the ability to pre-commit and choose from 3 different appointment slots by clicking directly on the email.
  Arms: Active choice; Financial incentive + Active choice
Behavioral: Financial incentive — The participant will receive the offering of $100 if s/he follows through with screening colonoscopy.
  Arms: Financial incentive + Active choice

SUMMARY:
This is an RCT aimed at testing different population-based approaches to increasing colorectal cancer screening through email outreach, including usual email communication, active choice, and active choice + financial incentive.

DETAILED DESCRIPTION:
This is an RCT aimed at testing different population-based approaches to increasing colorectal cancer screening. The investigators will randomize a cohort of employees between the ages of 50-64 to 3 arms of email communications: a.) Usual email communication; b.) Active choice- usual care + the ability to pre-commit directly through a web form; c.) Financial incentive- usual care + active choice + financial incentive for completion.

ELIGIBILITY:
Inclusion Criteria:

* Male and female employees of the University of Pennsylvania Health System who live within 30 miles of a health system endoscopy center.

Ages: 50 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2250 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Colonoscopy participation | 3 months
  The percentage of participants who follow through with screening colonoscopy.

SECONDARY OUTCOMES:
Email engagement | 3 months
  The percentage of participants who respond to the email (arm 2 and 3).
Scheduling of colonoscopy | 3 months
  The percentage of participants who schedule a procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Shivan Mehta, MD, Principal Investigator — University of Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mehta SJ, Feingold J, Vandertuyn M, Niewood T, Cox C, Doubeni CA, Volpp KG, Asch DA. Active Choice and Financial Incentives to Increase Rates of Screening Colonoscopy-A Randomized Controlled Trial. Gastroenterology. 2017 Nov;153(5):1227-1229.e2. doi: 10.1053/j.gastro.2017.07.015. Epub 2017 Jul 20. PMID 28734830